CLINICAL TRIAL: NCT00296205
Title: Phase II Trial of High-dose Cyclophosphamide for Moderate to Severe Refractory Multiple Sclerosis
Brief Title: Phase II High-Dose Cyclophosphamide for Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: I am changing locations to Johns Hopkins Medical Center
Sponsor: Stony Brook University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20055203
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2006-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cyclophosphamide; autoimmune
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide

SUMMARY:
The purpose of this study is to determine what percentage of patients receiving high-dose Cyclophosphamide may experience a halt in the worsening of their disease or experience improvement of their disease and for how long the benefit may last.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is the major disabling neurologic disease of young adults,and represents the most common immune-mediated inflammatory and demyelinating disorder of the central nervous system (CNS). Active inflammatory lesions contain components that include T cells, macrophages, and activated microglia. Within these lesions myelin is removed, axons are damaged and oligodendrocytes may be lost. In lesions undergoing inflammatory demyelination axonal injury also occurs. The disability MS produces is underscored by the nearly fifty percent of patients who will require ambulatory aids within 15 years after disease onset.

Currently, there is no cure for MS. Therapy is targeted at changing the short-term natural history of MS: to decrease attack rates and to postpone long-term disability. At present, interferon beta and glatiramer acetate form the foundation of therapy for relapsing MS. Mitoxantrone is approved for more severe cases of relapsing MS, such as those with rapidly accumulating neurologic impairments.

High-dose cyclophosphamide (HDC) is a non-bone marrow transplant treatment option for those afflicted by severe, refractory immune-mediated illnesses by pathologic autoreactive lymphocytes. The goal of this therapy is to induce immunoablation without myeloablation: that is, to eradicate offending B and T cells responsible for the illness while sparing the pluripotent blood stem cell of any ill effect. Since 1966, multiple publications on numerous immune-mediated illnesses have shown HDC without stem-cell rescue to decrease disease activity and improve quality of life

In this protocol we study HDC for severe, refractory MS. The primary goal is to assess the safety of HDC in this population, where no data exists regarding the tolerability of high-dose chemotherapy without stem-cell rescue. The treatment goal is not to induce disease regression (resolution of fixed neurologic deficits), but rather to stop disease progression without further remittive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of secondary progressive (SPMS), primary progressive (PPMS) or progressive relapsing (PRMS) multiple sclerosis
* A diagnosis of MS will be established by fulfilling criteria "Recommended Diagnostic Criteria for Multiple Sclerosis: Guidelines from the Internal Panel on the Diagnosis of Multiple Sclerosis"
* The subtype of MS will be established by the natural history of the disease
* Age >18 but < 75 years
* An extended disability status scale (EDSS) score of >3.5 after two standard treatment regimens IFNB1a IFNB1b Glatiramer acetate Mitoxanthrone Steroids, plasmapheresis or IVIG individually or in combination constitute a single treatment regimen
* Patient must have a left ventricular ejection fraction of > 45%
* Serum Creatinine <3mg/dL
* For women of childbearing potential, serum βHCG (less than seven days before start of cyclophosphamide)
* Willingness to participate in a clinical trial

Exclusion Criteria:

* Patients who are preterminal or moribund
* Patients with active malignancies
* Patients with chromosomal abnormalities or peripheral blood counts suggestive of myelodysplastic syndrome
* Patients with active bacterial or fungal infections requiring oral or intravenous antimicrobials are not eligible until resolution of the infection
* Pregnant women and breast-feeding women
* Patients with known intolerance to G-CSF

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2003-10; Study Completion 2006-02 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is to evaluate the response rate of MS patients after high-dose cyclophosphamide therapy as determined by a sustained (greater than 6 months) decrease of greater than or equal to 1.0 in their EDSS score.

SECONDARY OUTCOMES:
The secondary endpoint of this study is to evaluate time to EDSS score progression.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas E Gladstone, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

REFERENCES:
- [Result] Gladstone DE, Zamkoff KW, Krupp L, Peyster R, Sibony P, Christodoulou C, Locher E, Coyle PK. High-dose cyclophosphamide for moderate to severe refractory multiple sclerosis. Arch Neurol. 2006 Oct;63(10):1388-93. doi: 10.1001/archneur.63.10.noc60076. Epub 2006 Aug 14. PMID 16908728